CLINICAL TRIAL: NCT04318769
Title: An Affirmative Coping Skills Intervention to Improve Mental and Sexual Health of Sexual and Gender Minority Youth (AFFIRM): A Stepped Wedge Waitlist Crossover Trial
Brief Title: An Affirmative Coping Skills Intervention to Improve Mental and Sexual Health of Sexual and Gender Minority Youth
Acronym: AFFIRM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Shelley Craig, Professor, University of Toronto
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 35229
Record Dates: First submitted 2020-03-18; First posted 2020-03-24 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Mental Health Issue; Hiv; Stigma, Social; Coping Skills
Keywords: Sexual and gender minority youth; Cognitive behavioral therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Social Stigma; Coitus

STUDY DESIGN:
Intervention Model Description: Participants are allocated in a 2:1 fashion to arm 1: AFFIRM intervention; or arm 2: waitlisted control.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Participants are not blinded as they know which arm they are allocated too. Care providers and outcome assessors are blinded as the investigator runs the allocation sequence and outcomes are administered via survey weblink
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AFFIRM (Experimental): AFFIRM is an 8-session psychoeducational weekly group intervention
  Interventions: Behavioral: AFFIRM
- Waitlisted control (No Intervention): Waitlisted control

INTERVENTIONS:
Behavioral: AFFIRM — AFFIRM is an 8-session manualized group coping skills intervention focused on reducing sexual risk behaviours and psychosocial distress among SGMY. AFFIRM is delivered by two facilitators (primarily social workers and peers) through a combination of education and rehearsal (i.e., simulation of real-life experiences) in a manner that affirms participants' sexual and gender minority identities and experiences.
  Arms: AFFIRM

SUMMARY:
AFFIRM is an 8-session manualized group coping skills intervention focused on reducing sexual risk behaviours and psychosocial distress among SGMY. AFFIRM is delivered by two facilitators (primarily social workers and peers) through a combination of education and rehearsal (i.e., simulation of real-life experiences) in a manner that affirms participants' sexual and gender minority identities and experiences. AFFIRM is being tested in a five-year trial using a stepped wedge waitlist crossover design, where all participants receive the intervention in clusters.

DETAILED DESCRIPTION:
Session 1 focus

Introduction to cognitive behavioral therapy (CBT), exploring lesbian, gay, bisexual, transgender, and queer (LGBTQ)+ identities, and understanding minority stress.

Session 1 activities

Introductions

Discussing the theory and purpose of CBT approaches

Exploring stress and minority stress

Understanding the causes of stress in our lives

Session 2 focus

Understanding the impact of anti-LGBTQ attitudes and behaviors on stress.

Session 2 activities

Check in and review

Examining homophobia, heterosexism, and transphobia at the individual, institutional, and cultural level

Identifying how these experiences impact thoughts, feelings, and behaviors

Fostering strategies for both coping with and combating anti-LGBTQ discrimination at all levels

Session 3 focus

Understanding how thoughts impact feelings.

Session 3 activities

Check in and review

Distinguishing between thoughts and feelings

Exploring how thoughts influence feelings and behaviors

Identifying counterproductive thinking patterns

Recognizing negative self-talk and feelings of hopelessness

Learning thought stopping

Session 4 focus

Using thoughts to change feelings.

Session 4 activities

Check in and review

Increasing positive thinking and feelings of hope

Changing negative thoughts to positive thoughts

Challenging negative thinking and internalized homophobia/negative feelings through the ABCD (activating event, belief, consequence, and debate) method

Session 5 focus

Exploring how activities impact feelings.

Session 5 activities

Check in and review

Examining the impact of various activities on feelings

Identifying supportive and identity-affirming activities

The impact of LGBTQ-affirming activities on feelings

Session 6 focus

Planning to overcome counterproductive thoughts and negative feelings.

Session 6 activities

Check in and review

Distinguishing between clear and unclear goals

Identifying short, mid-, and long-term goals

Creating a sexual health plan

Fostering hope for the future

Session 7 focus

Understanding the impact of minority stress and anti-LGBTQ attitudes or behaviors on social relationships.

Session 7 activities

Check in and review

Anti-LGBTQ discrimination can lead to feelings of discomfort around others

Responding to discrimination or harassment in social situations

Learning to be assertive

Session 8 focus

Putting it all together: developing safe, supportive, and identity-affirming social networks.

Session 8 activities

Check in and review

Maintaining a healthy social network: attending to thoughts, expectations, feelings, and behaviors within relationships

Identifying a plan for building a supportive network

ELIGIBILITY:
Inclusion Criteria:

* Aged 14 to 29 years at time of screening
* Identifies as a sexual and/or gender minority
* Reads, writes, and speaks fluent English
* Is interested in participating in the 8-session AFFIRM intervention

Exclusion Criteria:

* Assessed to be in crisis (i.e., high risk of suicidality)
* Warrenting a more intensive intervention

Ages: 14 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Participants must self-identify as a sexual minority and/or as a gender minority
Enrollment: 300 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility - participant attendance at group sessions | week 56
  Proportions of participants that enroll, commence, and complete the intervention.
Acceptability - participant satisfaction with group sessions | week 56
  Participants will complete a satisfaction questionnaire.

SECONDARY OUTCOMES:
Intervention fidelity - how closely facilitators adhere to intervention model | Study period sessions 1-8 (weeks 1-8)
  Independent coders will complete a checklist questionnaire of AFFIRM intervention items, based on the manual, to determine how closely intervention facilitators adhered to the model

OTHER OUTCOMES:
Change in Sexual Health Capacity Scale | Baseline visit (week -1), postintervention visit (week 8), 6-month follow-up (week 32), 1-year follow-up (week 56)
  Four items. Scores range from 4 to 16. Higher scores mean better outcomes.
Abstinence Self-Efficacy Scale | Baseline visit (week -1), postintervention visit (week 8), 6-month follow-up (week 32), 1-year follow-up (week 56)
  Five items. Scores range from 5 to 20. Higher scores mean better outcomes.
Protection Self-Efficacy Scale | Baseline visit (week -1), postintervention visit (week 8), 6-month follow-up (week 32), 1-year follow-up (week 56)
  Eight items. Scores range from 8 to 32. Higher scores mean better outcomes
Change in DSM 5a Self-Rated Level 1 Cross-Cutting Symptom Measure - Child | Baseline visit (week -1), postintervention visit (week 8), 6-month follow-up (week 32), 1-year follow-up (week 56)
  Twenty items. Scores range from 0 to 80. Lower scores mean better outcomes.
Change in Current Mood Scale | Baseline visit (week -1), postintervention visit (week 8), 6-month follow-up (week 32), 1-year follow-up (week 56)
  Six items. Scores range from 0 to 60. Lower scores mean better outcomes.
Change in Beck Depression Inventory-II | Baseline visit (week -1), postintervention visit (week 8), 6-month follow-up (week 32), 1-year follow-up (week 56)
  Twenty items. Scores range from 0 to 80. Lower scores mean better outcomes.
Change in Brief COPE Scale | Baseline visit (week -1), postintervention visit (week 8), 6-month follow-up (week 32), 1-year follow-up (week 56)
  28 items. Scores range from 28 to 112. Higher scores mean better outcomes.
Change in Proactive Coping Inventory for Adolescents-A - Reflective Coping Subscale | Baseline visit (week -1), postintervention visit (week 8), 6-month follow-up (week 32), 1-year follow-up (week 56)
  11 items. Scores range from 0 to 33. Higher scores mean better outcomes.
Change in Stress Appraisal Measure for Adolescents | Baseline visit (week -1), postintervention visit (week 8), 6-month follow-up (week 32), 1-year follow-up (week 56)
  13 items. Scores range from 13 to 65. Higher scores mean better outcomes.
Change in Adult Hope Scale | Baseline visit (week -1), postintervention visit (week 8), 6-month follow-up (week 32), 1-year follow-up (week 56)
  12 items. Scores range from 12 to 96. Higher scores mean better outcomes.
Change in Internalized Homophobia Scale | Baseline visit (week -1), postintervention visit (week 8), 6-month follow-up (week 32), 1-year follow-up (week 56)
  10 items. Score range from 10 to 100. Lower scores mean better outcomes.
Change in Everyday Discrimination Scale | Baseline visit (week -1), postintervention visit (week 8), 6-month follow-up (week 32), 1-year follow-up (week 56)
  7 items. Scores range from 7 to 42. Higher scores mean better outcomes.
Change in LGBTQ Microaggressions Scale | Baseline visit (week -1), postintervention visit (week 8), 6-month follow-up (week 32), 1-year follow-up (week 56)
  15 items. Scores from 0 to 75. Lower scores mean better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Shelley L Craig, PhD, Principal Investigator — Professor
Locations (7):
- Canada (7):
  - COMPASS Health, Hamilton, Ontario
  - Hamilton Family Health Team, Hamilton, Ontario
  - Reach Out Centre for Kids - Positive Space Network, Oakville, Ontario
  - The 519 Church Street Community Centre, Toronto, Ontario
  - Sherbourne Health Centre, Toronto, Ontario
  - Asian Community AIDS Services (ACAS), Toronto, Ontario
  - Centre for Addiction and Mental Health (CAMH), Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available to other researchers.

REFERENCES:
- [Background] Craig SL, McInroy LB, Eaton AD, Iacono G, Leung VW, Austin A, Dobinson C. An Affirmative Coping Skills Intervention to Improve the Mental and Sexual Health of Sexual and Gender Minority Youth (Project Youth AFFIRM): Protocol for an Implementation Study. JMIR Res Protoc. 2019 Jun 6;8(6):e13462. doi: 10.2196/13462. PMID 31172957
- [Derived] Craig SL, Leung VWY, Hui JA, Iacono G, Pascoe RV, Dillon F, Austin A, Pang N, Dobinson C, Brooks AS. LGBTQ + Affirmative CBT: a hierarchical linear model of longitudinal outcomes and mechanisms of change. BMC Psychol. 2025 Sep 8;13(1):1006. doi: 10.1186/s40359-025-03314-7. PMID 40922004
- See also: Project Website — http://www.projectyouthaffirm.org